CLINICAL TRIAL: NCT01123954
Title: Evaluating the Safeness of Trivalent Subunit Inactivated Influenza Vaccines in Preventing Flu on Vietnamese Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: V71_21
Record Dates: First submitted 2010-03-24; First posted 2010-05-14 (Estimated); Last update posted 2011-12-14 (Estimated); Status verified 2011-12

CONDITIONS: Seasonal Influenza
Keywords: Seasonal influenza; Vaccine

ARMS (1):
- Arm 1 (Other)
  Interventions: Biological: Seasonal flu vaccine

INTERVENTIONS:
Biological: Seasonal flu vaccine — This phase II is performed as a monocenter study site in a population of healthy subjects aged 1 to 45 years. Enrolled subjects received one single IM dose of trivalent subunit inactivated influenza vaccine during the vaccination visit, according to the study protocol (follow-up period: 30 days)

SUMMARY:
The present study will evaluate the safety in healthy people aged 1- 45 years (male and female) after single intramuscular (IM) dose of trivalent subunit inactivated influenza vaccine till the 30-days follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy people with aged 1 to 45 years;
2. Previous history of not being vaccinated by any flu vaccines;
3. Women of childbearing potential agree to apply the contraceptive measures during the study period;
4. Do not have any acute or chronic diseases by screening;
5. Having the abilities of understanding and conforming the study plan;
6. Volunteer to the study;
7. Agree to vaccinate completely and conform the follow up procedure within 30 days after the first vaccination.

Exclusion Criteria:

1. Having the suspected symptoms of infecting flu: cough, sore throat, stuffy or running nose, headache, malaise, myalgia and arthralgia, weakness, chilly or sweat;
2. A prior history of allergy to any components of candidate vaccine;
3. Sensitive to eggs or chicken protein, kanamycin, neomycin sulphate, formaldehyde, cetyltrimethylammonium bromide (CTAB) and polysorbate 80;
4. Females who are pregnant or nursing (breastfeeding) mothers, or females of childbearing potential who are sexually active and have not used or do not plan to use acceptable birth control measures during the first 3 weeks after vaccination;
5. Being immuno deficiency due to treatment;
6. Using immunosuppressive drugs (belong to steroid group) within 06 months before vaccination;
7. Being sickness or cancer or HIV (+);
8. Participating in other study on drug or vaccination;
9. Receipt of other vaccine within 04 weeks before participating in the study;
10. Congenital malformation, mental disorder or members of family having the mental disorder;
11. Using immune globulin or blood products within 03 months before vaccination;
12. Having an acute or chronic diseases that can cause influence on the safety including: hepatic, renal, mental diseases or diabetes and transplantation;
13. Body temperature over 37.5 degree Celcius within 01 week before vaccination;
14. History of alcohol or drugs addicted within 05 years;
15. Planning to travel away from the study site among the visits.

Ages: 1 Year to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2010-01; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Using the single vaccination for volunteers and follow up within 30 days since the first vaccination to evaluate levels of safety (AEs) after vaccination | 30 days, including the follow-up period

CONTACTS AND LOCATIONS:
Locations (1):
- Department of examination and vaccination - Institute Pasteur of Ho Chi Minh City (LAM: Laboratoires d'Analysis Medicale), Ho Chi Minh City, Vietnam